CLINICAL TRIAL: NCT02340052
Title: Pain Map DK: a Prospective Cohort Study of Pain Treatment in 500 Hip Arthroplasty Patients at Different Danish Hospitals
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Anja Geisler, RCCN, Zealand University Hospital
Other Study IDs: SM1-AG-2014
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Postoperative Pain
Keywords: postoperative pain treatment
MeSH Terms: conditions — Pain, Postoperative | interventions — Analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Frederiksberg Hospital: 100 patients undergoing planned total hil arthroplasty
  Interventions: Drug: Pain treatment
- Koege hospital: 100 patients undergoing planned total hil arthroplasty
  Interventions: Drug: Pain treatment
- Naestved Hospital: 100 patients undergoing planned total hil arthroplasty
  Interventions: Drug: Pain treatment
- Hilleroed Hospital: 100 patients undergoing planned total hil arthroplasty
  Interventions: Drug: Pain treatment
- Nykoebing Falster Hospital: 100 patients undergoing planned total hil arthroplasty
  Interventions: Drug: Pain treatment

INTERVENTIONS:
Drug: Pain treatment — Registration af actual analgesic treatment and outcomes

SUMMARY:
This is a prospective observational cohorte study. The aim is to investigate actual pain treatment and outcomes in a large population of total hip arthroplasty patients at 5 different hospitals in Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Primary planned total hip arthroplasty, Able to understand and speak english or danish.

Exclusion Criteria:

* patients not able to cooperate, patients with alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Total hip arthroplasty patients
Sampling Method: Probability Sample
Enrollment: 501 (Actual)
Dates: Start 2014-04; Primary Completion 2016-05 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
NRS pain during mobilization | 6 hours postoperatively
Total morphine-eqv. opioid consumption | 24 hours postoperatively

SECONDARY OUTCOMES:
NRS pain at rest | 6 hours postoperatively
NRS pain at rest | 24 hours postoperatively
NRS pain during mobilization | 24 hours postoperatively
Nausea | 6 hours postoperatively
Nausea | 24 hours postoperatively
Vomiting | Number of episodes during 24 hours postoperatively
Dizziness | 6 hours postoperatively
Dizziness | 24 hours postoperatively
Sedation | 6 hours postoperatively
Sedation | 24 hours postoperatively
Length of hospital stay | Number of days until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD. PhD, Study Chair — Head of research, department of anaesthesiology, Koege hospital
Locations (3):
- Denmark (3):
  - Frederiksberg hospital, Frederiksberg, Sealand
  - Koege hospital, Koege, Sealand
  - Naestved hospital, Næstved, Sealand

REFERENCES:
- [Derived] Geisler A, Dahl JB, Thybo KH, Pedersen TH, Jorgensen ML, Hansen D, Schulze LK, Persson EI, Mathiesen O. Pain management after total hip arthroplasty at five different Danish hospitals: A prospective, observational cohort study of 501 patients. Acta Anaesthesiol Scand. 2019 Aug;63(7):923-930. doi: 10.1111/aas.13349. Epub 2019 Mar 18. PMID 30883668